CLINICAL TRIAL: NCT04216368
Title: Effect of Balance Training on Mobility and Activities of Daily Living in Sarcopenic Inpatients Aged 80+Years
Brief Title: Balance Trainning for Sarcopenic Inpatients Aged 80+ Years
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuxiang Liang (Other)
Responsible Party: Sponsor-Investigator, Yuxiang Liang, Physiotherapist, West China Hospital
Organization: West China Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019（596）
Record Dates: First submitted 2019-12-31; First posted 2020-01-02 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental)
  Interventions: Behavioral: balance training; Behavioral: resistance training
- controlled group (Other)
  Interventions: Behavioral: resistance training

INTERVENTIONS:
Behavioral: balance training — The training to improve balance is to work on the core muscle groups that help to maintain your posture.,and increase muscular strength.
  Arms: experimental group
Behavioral: resistance training — Resistance training is a form of exercise that improves muscular strength and endurance. During a resistance training workout, you move your limbs against resistance provided by your body weight, gravity, bands, weighted bars or dumbbells.

SUMMARY:
Resistance training and aerobic exercise have been recommended for sarcopenic patients. However, whether balance training would further benefit for sarcopenic patients on the basis of resistance training and aerobic exercise remains unclear. The purpose of this study is to explore the effect of balance training on improving the mobility of elderly patients with sarcopenia. Balance training involves doing exercises that strengthen the muscles that help keep the aged upright, including the legs and core. These kinds of exercises can improve stability and help prevent falls.

ELIGIBILITY:
Inclusion Criteria：

* Sarcopenia defined by the Asia Working Group of Sarcopenia (AWGS)
* Agree to participant this study and sign the informed consent
* Aged 80 years or over

Exclusion Criteria:

* Patients who could not follow the training plan due to cognitive impairment, emotional problems or any other reasons;
* Severe heart and lung diseases;
* Renal insufficiency;
* Any type of tumor;
* Bedridden patients

Ages: 80 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Fall rates | One year
  The incidence of falls during the first year of follow-up
The change of activities of daily living | 3 Months
  Basic activities of daily living (BADL) assessed by Barthel Index

SECONDARY OUTCOMES:
The change of usual gait speed | 3 months
The change of handgrip strength | 3 months
The change of the score of Short Physical Performance Battery | 3 Months
  The Short Physical Performance Battery (SPPB) is an objective assessment tool for evaluating lower extremity functioning in older persons.
The change of the score of Timed Up and Go test | 3 Months
  The Timed Up and Go test (TUG) is a simple test used to measure basic functional mobility and safety with mobility.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Yang, Study Director — West China Hospital; Jiaojiao Jiang, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital，Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided